CLINICAL TRIAL: NCT00375466
Title: Phase 4 Study of Tranexamic Acid for Elderly Patients Undergoing Combined Aortic Valve Replacement and Coronary Artery Bypass Surgery.
Brief Title: Tranexamic Acid, Hemorrhage and Transfusions After Combined Aortic Valve Replacement and Coronary Artery Bypass Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4.2006.1285; 2006-004561-34 (EudraCT Number)
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Hemorrhage
Keywords: Hemorrhage; Transfusion; Blood components; Fibrinolysis; Platelet activation
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (Experimental)
  Interventions: Drug: Tranexamic acid
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid 10 mg/kg as a bolus dose followed by an infusion of 1 mg/kg/hour. Bolus given before start of surgery, infusion continued during surgery.
  Other Names: Cykokapron ACT: B02A A02
  Arms: Tranexamic Acid
Drug: placebo — 0.9% sodium chloride 10 mg/kg, as a bolus injection before surgery followed by 1 mg/kg/h as an infusion during surgery
  Arms: placebo

SUMMARY:
In this study we will investigate whether tranexamic acid given as an intravenous bolus injection before start of surgery, followed by a continuous infusion during surgery reduces, perioperative hemostatic activation, and postoperative bleeding and the need for transfusions of blood components in elderly patients undergoing combined aortic valve replacement and coronary artery bypass surgery. Tranexamic acid will be compared with placebo (0.9% sodium chloride) in a randomized and double-blind study design.

The study hypothesis is that tranexamic acid will reduce hemostatic activation and postoperative hemorrhage and the need for blood component transfusions in this group of patients.

DETAILED DESCRIPTION:
It has previously been shown that elderly patients show signs of increased perioperative hemostatic activation after coronary artery bypass grafting. In particular, compared to younger patients, elderly patients had more extensive fibrinolysis postoperatively. The antifibrinolytic drug tranexamic acid has been shown to reduce fibrinolysis, bleeding, and the need for transfusions of blood components after various cardiac surgical procedures. In this study we will investigate whether tranexamic acid reduces perioperative activation of coagulation as measured by plasma concentrations of antithrombin, thrombin-antithrombin complex, and prothrombin fragment 1+2, whether tranexamic acid reduces perioperative fibrinolysis as measured by plasma concentrations of D-dimer, and whether tranexamic acid reduces platelet activation as measured by plasma concentrations of neutrophil activating peptide 2 and by flow cytometry in elderly (above 70 years of age) patients undergoing combined aortic valve replacement and coronary artery bypass surgery. The primary endpoint of the study will, however, be total postoperative bleeding and the need for transfusions of blood components during and after surgery. The need for transfusions will be registered during the whole hospital stay. Patients will be randomized into two groups and given either tranexamic acid or placebo (0.9% sodium chloride) as an intravenous bolus injection before start of surgery followed by an intravenous infusion during surgery. Blood samples for the above mentioned plasma concentration measurements will be drawn preoperatively, intraoperatively during CPB, and 30 minutes and 3, 5, and 20 hours postoperatively. Postoperative bleeding will be registered for 16 hours. The need for any transfusions of blood products will be registered for the whole hospital stay.

ELIGIBILITY:
Inclusion Criteria: Patients above 70 years of age scheduled for combined aortic valve replacement and coronary artery bypass surgery.

-

Exclusion Criteria: Patients younger than 70 years of age. Patients scheduled for other procedures than combined aortic valve replacement and coronary artery bypass surgery. Patients who are not treated with aspirin. Patients with a medical condition known to influence the hemostatic system. Patients treated with drugs other than aspirin during the last week before surgery that may influence the hemostatic system, such as warfarin (coumarin), non-steroidal antiinflammatory drugs, clopidogrel, heparin, low molecular heparins. Patients who are treated with systemic steroids. Patients with a serum creatinin concentration above 140 micromol/l. Patients with an INR above 1.5. Patients who are not able to give written informed concent.

-

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Transfusion of blood components | Intraoperatively and during postoperative stay

SECONDARY OUTCOMES:
Postoperative hemorrhage | First 16 hours postoperatively
Fibrinolysis | 20 hours postoperatively
Platelet activation | 20 hours postoperatively
Activation of coagulation | 20 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Pleym, MD, PhD, Study Chair — St. Olavs Hospital; Guri Greiff, MD, Principal Investigator — St. Olavs Hospital; Alexander Wahba, MD, PhD, Principal Investigator — St. Olavs Hospital; Roar Stenseth, MD, PhD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St. Olav University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Greiff G, Stenseth R, Wahba A, Videm V, Lydersen S, Irgens W, Bjella L, Pleym H. Tranexamic acid reduces blood transfusions in elderly patients undergoing combined aortic valve and coronary artery bypass graft surgery: a randomized controlled trial. J Cardiothorac Vasc Anesth. 2012 Apr;26(2):232-8. doi: 10.1053/j.jvca.2011.07.010. Epub 2011 Sep 15. PMID 21924636